CLINICAL TRIAL: NCT03058328
Title: Post-surgery Systemic Inflammation and Neuro-immune Interactions
Brief Title: The White Blood Cell Reactivity Following Surgical Trauma and Associated Regulatory Mechanisms.
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars I Eriksson, Professor, Senior Consultant, Karolinska University Hospital
Other Study IDs: POSINI2
Record Dates: First submitted 2017-01-13; First posted 2017-02-20 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Neuroinflammation
Keywords: Inflammation/physiopathology, Immune System/immunology,; Neuroimmunomodulation/physiology, General Surgery; Heart Rate/physiology*Vagus Nerve/physiology*
MeSH Terms: conditions — Neuroinflammatory Diseases; Inflammation | interventions — Neuropsychological Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whoole blood from which PBMCs (Peripheral Blood Monocytic Cells), plasma, serum will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive testing, testing of heart rate variability and blood samples — No intervention. Registration of ECG, cognitive testing and blood sampling is performed in the perioperative period and during follow up.

SUMMARY:
The purpose of this study is to describe numerical and functional changes in the white blood cell efter surgical trauma. Further, observed immune cell changes correlate to heart rate variability and cognitive function will be assessed.

DETAILED DESCRIPTION:
Surgical trauma causes release of damage-associated molecular patterns (DAMPs) and other alarmines (e.g. HMGB-1) targeting receptors on local cells of the innate immune system, such as macrophages. This cellular response to trauma is followed by a rapid release of an array of inflammatory mediators (e.g. TNFα, IL-1B, IL-6, IL-8, IL-10) being dependent on intracellular activation of nuclear factor NF-kB. Until recently it was believed that the brain is protected from this cascade of inflammatory mediators primarily due to an intact blood-brain-barrier (BBB). However, there is now a growing body of evidence that long term impairment of brain functions is associated with trauma-induced activation of the brain innate immune system with subsequent impairment of higher cognitive processes and risk for later permanent dementia. Yet, the link between systemic inflammation and cognitive impairment is not fully understood.

Recent studies have mapped periphery-to-brain-signaling after surgical trauma and the impact of major surgical trauma on the human brain by serial PET-imaging. In series of surgical patients, profound and biphasic changes in brain immune activity after surgery has been demonstrated after major abdominal surgery with signs of early depression followed by an increased immune activity at 3 months postoperatively. These biphasic changes in brain immunity seem to be aligned with simultaneous changes in whole blood immune reactivity to LPS suggesting a close link between brain and peripheral immune systems in regulation of acute inflammation and immune responses. Preclinical work in surgical animal models indicates disruption of the BBB with migration of peripheral macrophages into the brain as a pathway of potential importance. Evidence from an orthopedic surgery model in mice of trauma-induced altered hippocampal neuro-immune activity further raises the question whether peripheral markers of neurodegeneration (S100b, neurofilament light NFL, ptau, beta-amyloid) are associated with POCD.

The immune-regulatory role of the brain via the cholinergic anti-inflammatory reflex pathway (mediated by the vagal nerve) has been identified as potential target for immune-modulatory treatment strategies in systemic inflammation. We have moreover demonstrated a distinct release of human carotid body inflammatory mediators at hypoxia and gene expression related to inflammatory mediators, suggesting a potential role of the human carotid body in periphery-to-brain immune-signaling. Modulation of a vagal nerve-derived inflammatory reflex pathway by electrical stimulation has recently been successfully applied in treatment of chronic inflammation among patients with rheumatoid arthritis.

The hypothesis is that vagal nerve activity modulates systemic inflammation in patients after major surgery and that this modulation is associated with cognitive performance in the postoperative period.

With a more comprehensive understanding of immune-to-brain signaling after surgical trauma and how this biphasic inflammatory response pattern is regulated by cellular and neuronal components, the impact of immune modulation on key processes behind surgery-induced brain dysfunction can be explored, and possible neural and humoral targets for relevant anti-inflammatory treatments established.

In abdominal surgery patients we will map inflammatory periphery-to-brain communication by description of the temporal association between brain regulation of peripheral immunity (i.e., temporal changes in vagal nerve activity as measured by serial measurements of heart rate variability), repeated blood reactivity to LPS by serial ex vivo LPS challenge and simultaneous plasma/serum-borne CNS inflammatory and brain injury biomarkers to explore the impact of changes in systemic and brain immune function after surgery on long-term cognitive performance.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnosed prostate disease who are scheduled for elective robot assisted prostate surgery (RALP) and who are otherwise healthy
* A body mass index (BMI) below 33
* Mini-mental state examination (MMSE) scoring >23

EXCLUSION CRITERIA

Exclusion criteria are patients with:

* Neurodegenerative disease
* Significant psychiatric illness
* Previous stroke
* Pacemaker, myocardial infarction or cardiac arrhythmias,
* Known obstructive coronary artery disease, left ventricular hypertrophy or New York Heart Association (NYHA) class 2-4 heart failure
* Chronic pain or inflammatory disease such as rheumatoid arthritis, inflammatory bowel disease, SLE, psoriasis
* Steroidal therapy
* Statin medication
* Medication with ß-blockers, anti-cholinergic medication
* Poorly controlled diabetes mellitus or any other condition known to cause autonomic dysfunction
* Abuse of alcohol or drugs
* Previous splenectomy
* Presumed uncooperativeness or legal incapacity.

The patient should not have:

* undergone surgery the last 6 months
* been treated for cancer the last 12 months
* been treated for infectious disease the previous month.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Patients with diagnosed prostate disease who are scheduled for elective robot assisted prostate surgery (RALP) and who are otherwise healthy, with a BMI below 33 and who score >23 performance points on Mini-mental state examination (MMSE).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in subsets of Monocytes after surgical trauma | Up to 6 months after surgery
  Changes in subsets of Monocytes after surgical trauma

SECONDARY OUTCOMES:
T-cell numbers after surgical trauma. | Up to 6 months after surgery
  T-cell numbers after surgical trauma.
B-cell numbers after surgical trauma. | Up to 6 months after surgery
  B-cell numbers after surgical trauma.
T-cell functionality changes after surgical trauma. | Up to 6 months after surgery
  T-cell functionality changes after surgical trauma.
B-cell functionality changes after surgical trauma. | Up to 6 months after surgery
  B-cell functionality changes after surgical trauma.

OTHER OUTCOMES:
Genetic response to surgical trauma | Up to 6 months after surgery
  Genetic response to surgical trauma, i.e. white blood cell RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Lars I Eriksson, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden